CLINICAL TRIAL: NCT05534659
Title: Comparison of Benefit and Survival for Different Etiologies of Adult Patients With Hydrocephalus Between Programmable Cerebrospinal Fluid Ventricular Shunt and Non-programmable Cerebrospinal Fluid Ventricular Shunt
Brief Title: Comparison of Programmable and Non-programmable CSF Shunts Among Adult Hydrocephalus Patients With Different Etiologies
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202200775B0
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Hydrocephalus; Ventriculoperitoneal Shunt Malfunction
Keywords: Hydrocephalus; Programmable shunt; Long-term outcome
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Programmable valve(PV) group: Adult patients with hydrocephalus who received programmable ventricular CSF shunts operation.
  Interventions: Device: Programmable valve
- Non-programmable valve(NPV) group: Adult patients with hydrocephalus who received non-programmable ventricular CSF shunts operation.
  Interventions: Device: Non-programmable valve

INTERVENTIONS:
Device: Programmable valve — Programmable valve used in the study included Medtronic Strata, B-Braun ProGav, Codman Certas.
  Groups: Programmable valve(PV) group
Device: Non-programmable valve — Non-programmable valve used in the study was Medtronic CSF-flow control valve.
  Groups: Non-programmable valve(NPV) group

SUMMARY:
Programmable valve (PV) has been shown as a solution to the high revision rate in pediatric hydrocephalus patients, but it remains controversial among adults. This study is to compare the overall revision rate, revision cause, and revision-free survival between PV and non-programmable valve (NPV) in adult patients with different hydrocephalus etiologies.

DETAILED DESCRIPTION:
Relatively high revision rates up to 32% of CSF shunting operations remained an unsolved problem for neurosurgeons. The cause of revisions were diverse, including overdrainage/underdrainage, shunting system obstruction, infection or technical skill related. Programmable valve (PV) has been shown as a solution to the high revision rate in pediatric hydrocephalus patients, but it remains controversial among adults. This study is to compare the overall revision rate, revision cause, and revision-free survival between PV and non-programmable valve (NPV) in adult patients with different hydrocephalus etiologies.

The investigators reviewed the chart of all patients with hydrocephalus receiving index ventricular CSF shunt operations conducted at a single institution in northern Taiwan from January 2017 to December 2017. Patients included in the study were followed up for at least five years. Statistical tests including independent t-test, Chi-square test and Fisher's exact test were used for comparative analysis, and Kaplan-Meier curve using log-rank test was performed to compare the revision-free survival between the PV and NPV groups

ELIGIBILITY:
Inclusion Criteria:

* received shunting operations at Chang Gung Medical Foundation, Linkou Branch from 2017/01/01~2017/12/31

Exclusion Criteria:

* Patients who received index ventricular CSF shunt at other hospitals,
* Patients who received index ventricular CSF shunt before January 1st 2017,
* Patients who were younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who received CSF ventricular shunting operations at Chang Gung Medical Foundation, Linkou Branch, a tertiary medical center in northern Taiwan, would be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Initial Shunt revision rate | since the time of index operation until the initial revision or 2022/07/31
  the ratio of the total number of patients with at least one revision to the total number of patients included in this study
Total Shunt revision rate | since the time of index operation until the initial revision or 2022/07/31
  the ratio of the total number of revisions to the total number of ventricular CSF shunt operations
The cause of shunt revision | since the time of index operation until the initial revision or 2022/07/31
  the cause of the shunt malfunction warranting revision operation
Type of the revision operation | since the time of index operation until the initial revision or 2022/07/31
  the detailed description of the revision operation
Revision-free survival | since the time of index operation until the initial revision or 2022/07/31
  the interval between index operation and the initial revision

SECONDARY OUTCOMES:
Shunt revision-free survival among different hydrocephalus etiologies | since the time of index operation until the initial revision or 2022/07/31
  the individual interval between index operation and the initial revision among different hydrocephalus etiologies

CONTACTS AND LOCATIONS:
Overall Officials: ZHUO HAO Liu, PhD, Principal Investigator — Department of Neurosurgery Chang Gung Memorial Hospital Chang Gung Medical College and University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li M, Wang H, Ouyang Y, Yin M, Yin X. Efficacy and safety of programmable shunt valves for hydrocephalus: A meta-analysis. Int J Surg. 2017 Aug;44:139-146. doi: 10.1016/j.ijsu.2017.06.078. Epub 2017 Jun 22. PMID 28648796
- [Background] Rinaldo L, Bhargav AG, Nesvick CL, Lanzino G, Elder BD. Effect of fixed-setting versus programmable valve on incidence of shunt revision after ventricular shunting for idiopathic normal pressure hydrocephalus. J Neurosurg. 2019 Jun 7;133(2):564-572. doi: 10.3171/2019.3.JNS183077. Print 2020 Aug 1. PMID 31174190
- [Background] Reddy GK, Bollam P, Shi R, Guthikonda B, Nanda A. Management of adult hydrocephalus with ventriculoperitoneal shunts: long-term single-institution experience. Neurosurgery. 2011 Oct;69(4):774-80; discussion 780-1. doi: 10.1227/NEU.0b013e31821ffa9e. PMID 21508873